CLINICAL TRIAL: NCT03131882
Title: Comparing the Efficacy of Ultrasound Guided Hyaluronic Injection With Ultrasound Guided Corticosteroid Injection in Treatment of Trigger Finger
Brief Title: Efficacy of Ultrasound Guided Hyaluronic Injection in Treatment of Trigger Finger
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-58-04
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Trigger Digit
Keywords: trigger finger; trigger thumb; ultrasound guided; hyaluronic acid
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Hyaluronic Acid; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyaluronic acid (Experimental): Hyaluronic acid
  Interventions: Drug: Hyaluronic Acid
- Triamcinolone acetonide (Active Comparator): 10mg/ml Triamcinolone acetonide
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Hyaluronic Acid — 1 ml of Low molecular weight hyaluronic acid injection under ultrasound guidance after subcutaneous 0.5ml of 1%lidocaine injection
  Other Names: Hyalgan
  Arms: Hyaluronic acid
Drug: Triamcinolone Acetonide — 1ml of 10 mg of triamcinolone injection under ultrasound guidance after subcutaneous 0.5 ml 1%lidocaine injection
  Other Names: Shincort inj.
  Arms: Triamcinolone acetonide

SUMMARY:
Comparing the Efficacy of Ultrasound Guided Hyaluronic Injection with Ultrasound Guided Corticosteroid Injection in Treatment of Trigger Finger

DETAILED DESCRIPTION:
Randomized controlled trial which designed to compare the success rate, recurrence rate and functional outcomes of patients with trigger finger whom was treated with ultrasound guided hyaluronic acid injection to ultrasound guided corticosteroid injection

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years old
* Quinnell grade I, II, III
* Acute (< 6 months)

Exclusion Criteria:

* Quinnell grade IV
* Diabetes mellitus
* Rheumatoid arthritis
* Pregnancy
* Patient with prior injection or surgery of trigger finger
* Patient who are allergy to hyaluronic acid

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Success rate | 1 month, 3 month, 6 months
  reduction of symptom which needed no further treatment at follow up

SECONDARY OUTCOMES:
Pain score | 1 month, 3 month, 6 months
  Visual analogue scale changes
Functional outcome | 1 month, 3 months, 6 months
  Disability of the arm, shoulder and hand score

CONTACTS AND LOCATIONS:
Overall Officials: Thepparat Kanchanathepsak, M.D., Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of medicine Ramathibodi hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No